CLINICAL TRIAL: NCT06421194
Title: Functional and Nutritional Plant-based Mixed Protein Study (FuN Protein Study)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore Institute of Food and Biotechnology Innovation (Other Government)
Responsible Party: Principal Investigator, Melvin Leow, Principal Investigator, Singapore Institute of Food and Biotechnology Innovation
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2023/00944
Record Dates: First submitted 2024-05-09; First posted 2024-05-20 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: Nutrition, Healthy
Keywords: plant-based protein; Asian; diet; health outcomes; animal-based protein

STUDY DESIGN:
Intervention Model Description: A randomized controlled crossover trial, where participants will undergo four sessions, each followed by a six-day wash-out period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Treatment 1 Animal-based protein meal (Experimental): Animal-based protein meal; Isoproteic at ~30g of total protein per meal. Siew mai (6 pieces) - steamed Ngoh Hiang (2 pieces) - oven baked
  Interventions: Other: Investigational meal 1 - Commercial animal-based protein foods [Siew mai (6 pieces) and Ngoh hiang (2 pieces)]
- Treatment 2 Animal-based protein meal (Experimental): Animal-based protein meal; Isoproteic at ~30g of total protein per meal. Gyoza (11 pieces) - steamed Luncheon meat (5 pieces) - oven baked
  Interventions: Other: Investigational meal 2- Commercial animal-based protein foods [Gyoza (11 pieces) and Luncheon meat (5 pieces)]
- Treatment 3 Plant-based protein meal (Experimental): Plant-based protein meal; Isoproteic at ~30g of total protein per meal. Siew mai (6 pieces) - steamed Ngoh Hiang (1 piece cut into 2) - oven baked
  Interventions: Other: Investigational meal 3- Formulated plant-based protein foods [Siew mai (6 pieces) and Ngoh hiang (1 piece cut into 2)]
- Treatment 4 Plant-based protein meal (Experimental): Plant-based protein meal; Isoproteic at ~30g of total protein per meal. Gyoza (11 pieces) - steamed Luncheon meat (5 pieces) - oven baked
  Interventions: Other: Investigational meal 4- Formulated plant-based protein foods [Gyoza (11 pieces) and Luncheon meat (5 pieces)]

INTERVENTIONS:
Other: Investigational meal 1 - Commercial animal-based protein foods [Siew mai (6 pieces) and Ngoh hiang (2 pieces)] — Participants consume a meal consisting of commercial animal-based protein foods (steamed Siew mai and oven-baked Ngoh hiang) in a fasted state.
  Arms: Treatment 1 Animal-based protein meal
Other: Investigational meal 2- Commercial animal-based protein foods [Gyoza (11 pieces) and Luncheon meat (5 pieces)] — Participants consume a meal consisting of commercial animal-based protein foods (steamed Gyoza and oven-baked Luncheon meat) in a fasted state.
  Arms: Treatment 2 Animal-based protein meal
Other: Investigational meal 3- Formulated plant-based protein foods [Siew mai (6 pieces) and Ngoh hiang (1 piece cut into 2)] — Participants consume a meal consisting of formulated plant-based protein foods (steamed Siew mai and oven-baked Ngoh hiang) in a fasted state.
  Arms: Treatment 3 Plant-based protein meal
Other: Investigational meal 4- Formulated plant-based protein foods [Gyoza (11 pieces) and Luncheon meat (5 pieces)] — Participants consume a meal consisting of formulated plant-based protein foods (Gyoza and Luncheon meat) in a fasted state.
  Arms: Treatment 4 Plant-based protein meal

SUMMARY:
The study aims to investigate the effects of optimized plant protein mixtures versus their animal protein equivalents on satiety, protein metabolism, and overall metabolic health

DETAILED DESCRIPTION:
The research described in this application is crucial as it addresses a fundamental issue - the nutrition quality of plant-based diets. Plant-based diets are widely acknowledged for their health benefits as they are known to reduce disease risks and all-cause mortality. However, concerns about plant protein quality arise due to disparities in amino acid profiles, particularly their essential amino acid adequacy, which remains a challenge in adopting a plant-based protein diet as part of a healthy diet. Other challenges include low palatability, poor texture, flavor, and mouthfeel. To address this, the Singapore Institute of Food and Biotechnology Innovation (SIFBI) has developed Asian-centric plant-based food products by combining multiple plant-protein sources to emulate the amino acid profile of animal proteins. This approach aims to optimize plant-based diets by ensuring enhanced protein quantity and quality in a mixed meal, not only to encourage adaptation of plant based protein into daily meals for environmental sustainability but also with the long-term objectives to use diet as a means to improve metabolic health in the Asian demographics. This human study is designed to explore the effects of consuming optimized plant-protein-based products compared to conventional animal protein- based products on postprandial metabolism and overall metabolic health. The study is structured around several specific objectives:

1. Evaluate Nutritional Impact: The study aims to assess the nutritional efficacy of the investigational food products. This will involve measuring circulating amino acids and protein metabolism markers, such as blood urea and amino acid metabolites. Additionally, the study will examine the effects of these foods on overall metabolic health, including their impact on glycaemic response and inflammatory markers.
2. Investigate Postprandial Satiety: Another key aim is to explore the effects of investigational food items on postprandial appetite and satiety. This will help determine how these foods influence hunger and fullness sensations following consumption, which is crucial for understanding their potential role in weight management and metabolic regulation.
3. Investigate Consumer Acceptance: The study will also assess consumer acceptance of the investigational food products to identify the potential barriers. This includes evaluating the palatability of these products, as their taste, texture, and overall appeal are vital factors in determining their potential integration into regular diets.
4. Gain Mechanistic Insight: The study seeks to gain deeper mechanistic insights by systematically investigating changes in the postprandial circulating proteome. This analysis will enhance our understanding of the biological processes and pathways involved in the body's response to these food products post-consumption.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Chinese ethnicity
* Age between 21 to 45 years
* Body Mass Index (BMI) between 18.5 to 27.5 kg/m2
* English-literate

Exclusion criteria:

* Smoking
* Having allergies or intolerances to any common food ingredients including eggs, fish, milk, peanuts, and tree nuts, shellfish, soya, wheat, pea, gluten, cereal, fruits, dairy products, meat, vegetable, sugar and sweetener, natural food colourings or flavourings, etc.
* Following special diets or having intentional dietary restrictions (e.g., vegetarians/vegans)
* Having a dislike towards plant-based or chicken-based foods
* Not willing to adhere to diet modification as in the study's instructions
* Not willing to stop any strenuous activity during or within 24 hours of test days
* Having glucose-6-phosphate dehydrogenase deficiency (G6PD deficiency)
* Having alcohol consumption on > 4 days per week with ≥ 6 alcoholic drinks per week
* Having sustained elevation of blood pressure (>160/95 mm Hg)
* HbA1c reading ≥ 6.5% (raised non-fasted/random HbA1c as defined by WHO/ IDF)
* Having previously undergone any gastrointestinal surgery or having history of gastrointestinal disorders
* Having a history of heart, liver, kidney, blood disorders (e.g., thalassemia) or thyroid dysfunctions
* Diabetic
* Having history of tuberculosis, HIV, Hepatitis B or Hepatitis C infections
* Having any prescription medication or any other alternative medicines or supplements (amino acids supplements, e.g. L-carnitine, glutamine and arginine) which may interfere with study measurements in the opinion of the study investigators
* Having antibiotics or suffering from diarrhoea within the last 4 weeks
* Having donated blood within 4 weeks of study participation
* Having poor veins or having history of severe vasovagal syncope (blackouts or fainting) from blood draws
* Employees of the SIFBI (Singapore Institute of Food and Biotechnology Innovation).

Ages: 21 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 28 (Estimated)
Dates: Start 2024-02-23 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Free amino acids | The initial baseline (before investigational meal) at 0 minute, and eight intervals post-meal at 15, 30, 45, 60, 90, 120, 150, and 180 minutes.
  Blood samples collected at 0, 15, 30, 45, 60, 90, 120, 150 and 180 minutes (plasma and serum)
Protein utilization | The initial baseline (before investigational meal) at 0 minute, and eight intervals post-meal at 15, 30, 45, 60, 90, 120, 150, and 180 minutes.
  Blood samples collected at 0, 15, 30, 45, 60, 90, 120, 150 and 180 minutes (plasma and serum)
Glucose homeostasis | The initial baseline (before investigational meal) at 0 minute, and eight intervals post-meal at 15, 30, 45, 60, 90, 120, 150, and 180 minutes.
  Blood samples collected at 0, 15, 30, 45, 60, 90, 120, 150 and 180 minutes (serum)
Gut hormones | The initial baseline (before investigational meal) at 0 minute, and eight intervals post-meal at 15, 30, 45, 60, 90, 120, 150, and 180 minutes.
  Blood samples collected at 0, 15, 30, 45, 60, 90, 120, 150 and 180 minutes (plasma and serum)
Markers related to general metabolic health | The initial baseline (before investigational meal) at 0 minute, and eight intervals post-meal at 15, 30, 45, 60, 90, 120, 150, and 180 minutes.
  Blood samples collected at 0, 15, 30, 45, 60, 90, 120, 150 and 180 minutes (plasma and serum)

SECONDARY OUTCOMES:
Untargeted proteomics | The initial baseline (before investigational meal) at 0 minute, and eight intervals post-meal at 15, 30, 45, 60, 90, 120, 150, and 180 minutes.
  To study molecular mechanism underlying the observed outcomes (plasma and serum).
Visual Analogue Scale Questionnaire | The initial baseline (before investigational meal) at 0 minute, and eight intervals post-meal at 15, 30, 45, 60, 90, 120, 150, and 180 minutes.
  To assess participant's postprandial appetite and satiety, participants complete, C a Visual Analogue Scale (VAS) questionnaire pertaining to their appetite.
  At baseline time 0 minute, one question will be asked and participants will mark on a scale to indicate how they feel at that moment.
  A. Questions on appetite and desire for specific food type (how hungry you feel, how satisfied you feel, how full you feel, how much do you think you can eat)
  Time 15 minute to time 180 minute (8 time points, post meal), following two questions will be asked and participants will mark on a scale to indicate how they feel at that moment.
  A. Questions on appetite and desire for specific food type (how hungry you feel, how satisfied you feel, how full you feel, how much do you think you can eat) B. Questions on palatability of test meal (to complete immediately after meal intake) (visual appeal, smell, taste, aftertaste, palatibility)
Gastrointestinal Symptoms Questionnaire | The initial baseline (before investigational meal) at 0 minute, and eight intervals post-meal at 15, 30, 45, 60, 90, 120, 150, and 180 minutes.
  Participants complete a questionnaire pertaining to their gastrointestinal (GI) symptoms before investigational meal (0 minute) and at the end of the session (180 minute). Gastrointestinal symptoms pertaining to flatulence, rumbling, bloating, abdominal pain, abdominal cramps, nausea.

CONTACTS AND LOCATIONS:
Overall Officials: Melvin Leow, Professor, Principal Investigator — Singapore Institute of Food and Biotechnology Innovation (SIFBI), A*STAR
Locations (1):
- Clinical Nutrition Research Centre, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No